CLINICAL TRIAL: NCT01747538
Title: A Randomized, Double-masked, Placebo-controlled Study of the Safety and Efficacy of Gevokizumab in the Treatment of Subjects With Non-infectious Intermediate, Posterior, or Pan-uveitis Currently Controlled With Systemic Treatment
Brief Title: Safety and Efficacy Study of Gevokizumab to Treat Non-infectious Uveitis Controlled With Systemic Treatment
Acronym: EYEGUARD™-C
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Collaborators: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X052131/CL3-78989-006; 2012-001609-25 (EudraCT Number); U1111-1135-1462 (Other: WHO)
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Uveitis
Keywords: Uveitis; Non-infectious Uveitis; Intermediate Uveitis; Posterior Uveitis; Panuveitis
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Uveitis, Posterior; Panuveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dose 1 gevokizumab (Experimental)
  Interventions: Drug: Dose 1 gevokizumab
- Dose 2 gevokizumab (Experimental)
  Interventions: Drug: Dose 2 gevokizumab

INTERVENTIONS:
Drug: Placebo — Solution for subcutaneous injection
  Arms: Placebo
Drug: Dose 1 gevokizumab — Solution for subcutaneous injection
  Arms: Dose 1 gevokizumab
Drug: Dose 2 gevokizumab — Solution for subcutaneous injection
  Arms: Dose 2 gevokizumab

SUMMARY:
The purpose of this study is to evaluate the efficacy of gevokizumab in reducing the risk of recurrent uveitic disease in subjects with non-infectious uveitis whose disease is currently controlled with systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-infectious intermediate, posterior, or pan- uveitis in at least one eye
* Controlled uveitic disease in both eyes
* Stable dose of oral corticosteroids in combination with selected stable immunosuppressive therapy
* Effective contraceptive measures

Exclusion Criteria:

* Infectious uveitis and masquerade syndromes
* Isolated anterior uveitis
* Contraindication to mydriatics
* Active tuberculosis disease
* History of allergic or anaphylactic reactions to monoclonal antibodies
* History of recurrent infection or predisposition to infection; active ocular infection
* Pregnant or nursing women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an occurrence of uveitic disease through Day 168 | Day 0 through Day 168

SECONDARY OUTCOMES:
Time to first occurrence of uveitic disease | Day 0 through Day 168

CONTACTS AND LOCATIONS:
Locations (114):
- United States (51):
  - Chandler, Arizona
  - Phoenix, Arizona
  - Beverly Hills, California
  - Los Angeles, California
  - Redlands, California
  - Sacramento, California
  - San Luis Obispo, California
  - Santa Ana, California
  - Victorville, California
  - Golden, Colorado
  - Littleton, Colorado
  - Bridgeport, Connecticut
  - Washington D.C., District of Columbia
  - Lakeland, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Ellsworth, Maine
  - Baltimore, Maryland
  - Cambridge, Massachusetts
  - Waltham, Massachusetts
  - Detroit, Michigan
  - Jackson, Michigan
  - Royal Oak, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Bloomfield, New Jersey
  - Palisades Park, New Jersey
  - Teaneck, New Jersey
  - Belmont, North Carolina
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Beachwood, Ohio
  - Cleveland, Ohio
  - Middleburg Heights, Ohio
  - Ashland, Oregon
  - Philadelphia, Pennsylvania
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Mission, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
- Argentina (3):
  - Olivos, Buenos Aires
  - Rosaria, Santa Fe Province
  - Buenos Aires
- Yerevan, Armenia
- Australia (4):
  - Sydney, New South Wales
  - East Melbourne, Victoria
  - Nedlands, Western Australia
  - Darlinghurst, New South Wales
- Brazil (3):
  - Belo Horizonte, Minas Gerais
  - Rio de Janeiro
  - São Paulo
- Canada (2):
  - Ottawa, Ontario
  - Montreal, Quebec
- China (3):
  - Beijing
  - Chongqing
  - Hong Kong
- France (3):
  - Lyon
  - Nantes
  - Paris
- Germany (5):
  - Berlin
  - Chemnitz
  - Heidelberg
  - Münster
  - Tüebingen
- Mezourlo, Larissa, Greece
- Israel (3):
  - Jerusalem
  - Petoch Tikvah
  - Tel Aviv
- Italy (5):
  - Ancona, Marche
  - Genova
  - Milan
  - Padua
  - Romagna
- Mexico (4):
  - Distrito Federal
  - Mexico City
  - Nuevo León
  - Tijuana
- Poland (4):
  - Gdansk
  - Katowice
  - Lublin
  - Warsaw
- Portugal (3):
  - Braga
  - Coimbra
  - Lisbon
- Russia (3):
  - Khabarovsk
  - Novosibirsk
  - Saint Petersburg
- South Africa (2):
  - Durban
  - Johannesburg, Gauteng
- Spain (4):
  - Barcelona
  - Granada
  - Madrid
  - Málaga
- Taiwan (2):
  - Taïpeï City
  - Taoyuan District
- Monastir, Tunisia
- Turkey (Türkiye) (3):
  - Ankara
  - Cerrahpasa, Istanbul
  - Faith, Istanbul
- United Kingdom (4):
  - Sunderland, Tyne and Wear
  - Bristol
  - Liverpool
  - London